CLINICAL TRIAL: NCT01172496
Title: A Comparative Bioavailability Study of UT-15C SR (Treprostinil Diethanolamine, Sustained Release) Oral Tablets and UT-15C (Treprostinil Diethanolamine) Administered as an Oral Solution in Healthy Volunteers
Brief Title: A Bioavailability Study Comparing Treprostinil Diethanolamine Oral Tablets and Oral Solution in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Kevin Laliberte, PharmD; Senior Director, Product Development, United Therapeutics
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TDE-PH-123
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-07

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

ARMS (2):
- 1 mg tablet; 1mg solution (Experimental)
  Interventions: Drug: treprostinil diethanolamine
- 1mg solution; 1mg tablet (Experimental)
  Interventions: Drug: treprostinil diethanolamine

INTERVENTIONS:
Drug: treprostinil diethanolamine — Subjects will be administered a 1 mg dose of treprostinil diethanolamine as a single tablet, and treprostinil diethanolamine oral solution 0.25 mg dose every 2 hours for four doses (1 mg total).

SUMMARY:
This single center, open label, randomized, two-period, two-sequence cross-over study is designed to evaluate the relative bioavailability of a treprostinil diethanolamine 1 mg tablet in reference to treprostinil diethanolamine 1 mg oral solution (administered as four 0.25 mg doses every 2 hours for a 1 mg total dose) in twenty-four healthy volunteers. Other secondary outcomes of interest include assessment of pharmacokinetic parameters of treprostinil diethanolamine 1 mg tablets and a treprostinil diethanolamine 1 mg oral solution administered as four doses (0.25 mg every 2 hours for a 1 mg total dose) and evaluation of the safety and tolerability of each treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy between the ages of 18-55 years of age
* Female subjects must weigh between 55 and 100 kg, with a BMI between 19.0-29.9. kg/m2; inclusive at screening. Male subjects must weigh between 55 and 120 kg, with a BMI between 19.0-32.0 kg/m2; inclusive at screening.
* Subject has a medical history, physical examination, vital signs, ECG and clinical laboratory results within normal limits or considered not clinically significant by the Investigator at Screening.
* Female subjects with childbearing potential will practice abstinence or effective birth control methods from the time of providing written informed consent to the end of the study. Effective birth control is defined as an intrauterine device (IUD), barrier methods preferably in combination with a spermicidal foam or suppository, or the use of oral, transdermal or intra-vaginal hormonal contraceptives.
* Subject agrees to abstain from taking any prescription medication (except contraceptives) for 14 days prior to starting study procedures and to abstain from taking any non-prescription medications (except multivitamins) or herbal supplements for 7 days prior to beginning study procedures until discharge from the study (unless prescribed by the Investigator to treat an AE).
* Subject agrees to abstain from consuming alcohol from 3 days prior beginning study procedures until discharge from the study.
* Subject agrees to abstain from consuming grapefruit or xanthine-containing food or beverages for 3 days prior beginning study procedures until discharge from the study.
* Subject agrees to refrain from strenuous exercise from beginning study procedures until discharge from the study.
* Subject is able to communicate effectively with study personnel and be considered reliable, willing and cooperative in terms of compliance with the protocol requirements.

Exclusion Criteria:

* Subject has any clinically relevant abnormality identified during the screening physical examination, 12-lead ECG, or laboratory examinations.
* Subject has a history of anaphylaxis, a previous documented hypersensitivity reaction, or a clinically significant idiosyncratic reaction to any drug.
* Subject has a clinically significant history of neurological, cardiovascular, respiratory, endocrine, hematological, hepatic, renal, gastrointestinal, genitourinary, pulmonary, and/or musculoskeletal disease; glaucoma; a psychiatric disorder, or any other chronic disease, whether controlled by medication or not.
* The subject has a history of postural hypotension, unexplained syncope, a blood pressure that is less than 85 mmHg systolic or 50 mmHg diastolic, or a pulse rate that is greater than 90 bpm after sitting at rest for 5 minutes at Screening or Baseline.
* Subject has a predisposing condition that could interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Subject has tested positive at the screening visit for HIV infection, HBsAg, or the HCV antibody.
* Subject is pregnant or lactating.
* Subject currently uses tobacco products or has a history of tobacco use within six months prior to Period 1.
* Subject has a history of alcohol abuse or a history of or current impairment of organ function reasonably related to alcohol abuse.
* Subject has a history of or current evidence of abuse of licit or illicit drugs or a positive urine screen for drugs of abuse.
* Subject has a history of abnormal bleeding tendencies.
* Subject has donated blood or plasma or has lost a significant volume of blood (greater than 450 mL) within four weeks prior to Period 1.
* Subject has participated in any investigational drug study within 30 days prior to Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Plasma treprostinil concentrations | 1 month
  Pharmacokinetic blood sampling will occur twice for each subject. Pharmacokinetic parameters will be derived from treprostinil concentration-time data

SECONDARY OUTCOMES:
vital sign measurements, clinical laboratory parameters, electrocardiograms (ECGs) and adverse events (AEs) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Laurent, MD, Principal Investigator — PPD Development, LP
Locations (1):
- PPD Development, Austin, Texas, United States